CLINICAL TRIAL: NCT02115763
Title: The Effects of Caffeine on Pain-Based Pacing During a Cycling Time-Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 4084
Record Dates: First submitted 2014-04-11; First posted 2014-04-16 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Healthy
Keywords: physically active,; 18-35 year old men
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Caffeine (Experimental): There is only one arm, it receives both caffeine and placebo.
  Interventions: Drug: Caffeine; Drug: Placebo

INTERVENTIONS:
Drug: Caffeine
Drug: Placebo

SUMMARY:
Caffeine has been shown to consistently improve time-trial performance, warranting restrictions on consumption under regulation of the National Collegiate Athletics Association (NCAA) and World Anti-Doping Agency (WADA). This ergogenic effect is not well understood, possibly occurring as a result of altered metabolism, improved strength, and/or reduced muscle pain. The hypothesis of altered metabolism has recently fallen out of favor while muscular strength has a tenuous relationship with endurance exercise performance. Reductions in muscle pain have been observed during low and moderate intensity endurance exercise, and this may be the mechanism of caffeine's ergogenic effect. In lieu of reducing pain during high intensity exercise, caffeine significantly improves performance. Therefore, caffeine appears to improve the amount of work that can be done for a given muscle pain rating, suggesting that participants may pace based upon sensations of muscle pain during endurance exercise. Most time-trial exercise is conducted in a fixed distance manner, measuring the time it takes participants to cover a given distance. Little research has been conducted on a fixed pain time-trial that would require participants to produce and sustain a given level of muscle pain while measuring the distance covered in an allotted time. A fixed pain time-trial could allow researchers to better understand the effect of pain on endurance performance. The purpose of this study is to examine the effects of caffeine on a fixed pain time-trial.

ELIGIBILITY:
Inclusion Criteria:

* Caffeine Naive (<40mg per day) physically active 18-35 year old men with no contraindications to exercise.

Exclusion Criteria:

* People who do not match the gender, age or caffeine limits;
* those with contraindications to exercise or who are not physically active

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Stationary Cycle Ergometer | 30 minutes per session (6 sessions total)
  The distance covered (meters) while exercising on the cycle ergometer will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oklahoma Sensory and Muscle Function Lab, Norman, Oklahoma, United States